CLINICAL TRIAL: NCT04267575
Title: Canady Helios Cold Plasma Scalpel Treatment at the Surgical Margin and Macroscopic Tumor Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jerome Canady, M.D. (Other)
Responsible Party: Sponsor-Investigator, Jerome Canady, M.D., Sponsor-Investigator, Jerome Canady Research Institute for Advanced Biological & Technological Sciences
Organization: Jerome Canady Research Institute for Advanced Biological & Technological Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G190165
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Recurrent Malignant Solid Neoplasm; Stage IV Breast Cancer; Stage IV Prostate Cancer; Stage IV Pancreatic Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Cancer; Stage IV Fallopian Tube Cancer; Stage IV Colon Cancer; Stage IV Colorectal Cancer; Stage IV Liver Cancer; Stage IV Renal Cell Cancer; Stage IV Rectal Cancer; Stage IV Lung Cancer; Stage IV Small Intestinal Cancer; Stage IV Gastric Cancer; Stage IV Bladder Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Fallopian Tube Neoplasms; Colonic Neoplasms; Colorectal Neoplasms; Liver Neoplasms; Carcinoma, Renal Cell; Rectal Neoplasms; Lung Neoplasms; Stomach Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Primary Arm (Experimental): After the gross solid tumor is removed, cold plasma is sprayed in the area of the resected tumor margins.
  Interventions: Device: Canady Helios Cold Plasma Scalpel

INTERVENTIONS:
Device: Canady Helios Cold Plasma Scalpel — Device used to distribute cold plasma energy at the resected tumor margins.

SUMMARY:
The study designed is to evaluate the safety of Canady Helios™ Cold Plasma Scalpel (CHCPS) in patients with solid tumors with carcinomatosis scheduled to undergo surgical resection for cytoreduction. Patients with stage 4 resectable tumors as decided by a multidisciplinary disease management team may be included if the metastatic disease is non-synchronous (e.g. recurrent colorectal carcinoma with hepatic metastasis amenable for surgical resection).. Plasma is an ionized gas typically generated in high-temperature laboratory conditions. Plasma coagulators are currently used routinely as surgical tools with multiple applications that create temperatures between 37° C to 43°C and cause thermal injury. Earlier studies demonstrated the non-aggressive nature of cold plasma. As evidence accumulates, it is becoming clear that low-temperature cold plasma has an increasing role in biomedical applications.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Solid tumors undergoing surgical treatment with carcinomatosis scheduled to undergo surgical resection for cytoreduction. Patients with stage 4 resectable tumors as decided by a multidisciplinary disease management team may be included if the metastatic disease is non-synchronous (e.g. recurrent colorectal carcinoma with hepatic metastasis amenable for surgical resection).
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study and must be willing to return for follow-up
* 18 years of age or older and capable of providing informed consent indicating awareness of the investigational nature of this trial, in keeping with Good Clinical Practice (GCP) guidelines and institutional policy.
* Biopsy (histopathology or cytology) diagnosis of a solid tumor as defined by the World Health Organization (WHO) or by cross-sectional imaging reviewed by a board-certified radiologist.
* Good performance status (ECOG < 2), Karnofsky >60%,
* Patients with low or acceptable surgical risk (American society of Anesthesiology (ASA) score of 3 or less.
* Patient is a candidate for surgical therapy as discussed and recommended by the institutional disease management team (DMT, Tumor Board).

At the time of enrollment:

* Absolute neutrophil count (ANC) exceeds 1200/mm3, white blood cell count exceeds 4000/mm3 and platelet count is greater than 100,000/mm3
* An international normalized ratio (INR) ≤ 1.5 (patients who are therapeutically anticoagulated for non-related medical conditions such as atrial fibrillation and whose anti-thrombotic treatment can be withheld for operation will be eligible).
* Adequate hepatic function must be met as evidenced by total serum bilirubin ≤ 3.0 mg/dl ; alkaline phosphatase < 2.5 times the upper limit of normal; and, aspartate aminotransferase (AST) less than 1.5 times upper limit of normal [alkaline phosphatase and AST cannot both exceed the upper limit of normal]
* Serum renal functional parameters, blood urea nitrogen (BUN) and creatinine are within normal limits
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
* Life expectancy of at least six months

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patients with unresectable tumors as decided by a multidisciplinary disease management team
* Patients with multiple metastatic sites not amenable for surgical resection
* Pregnancy or lactation
* Patients with low performance status (ECOG > 2 or Karnofsky < 60%)
* Any one or more of the following hematological abnormalities
* Hgb < 8gm/dl unable to be corrected with transfusion
* Absolute Neutrophil Count < 1200/mm3
* White blood cell count < 4000/mm3
* Platelet count < 100,000/mm3
* INR > 1.5 (except in patients who are therapeutically AST anticoagulated for non-related medical conditions such as atrial fibrillation and whose anti-thrombotic treatment cannot be withheld for operation will be eligible)
* History of hepatic cirrhosis or present hepatic dysfunction
* Alkaline phosphatase ≥ 2.5 times the upper limit of normal
* ≥ 1.5 times upper limit of normal
* Serum bilirubin > 3.0 mg/dl
* Alkaline phosphatase and AST both exceed the upper limit of normal
* Renal insufficiency indicated by a serum creatinine >1.5mg/dL.
* Patients with high surgical risk (ASA 4-5) with significant history of a medical problem that would preclude the patient from undergoing an operative procedure such as a history of severe congestive heart failure or active ischemic heart disease.
* Febrile illness within 7 days before scheduled surgery
* Treatment with another investigational drug or other intervention within 60 days before surgery
* Patients that are unable to- or unwilling to provide a written informed consent
* Patients who underwent treatment with cold plasma within a year before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2023-04-14 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Canady Surgical Group PC, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Canady J, Murthy SRK, Zhuang T, Gitelis S, Nissan A, Ly L, Jones OZ, Cheng X, Adileh M, Blank AT, Colman MW, Millikan K, O'Donoghue C, Stenson KM, Ohara K, Schtrechman G, Keidar M, Basadonna G. The First Cold Atmospheric Plasma Phase I Clinical Trial for the Treatment of Advanced Solid Tumors: A Novel Treatment Arm for Cancer. Cancers (Basel). 2023 Jul 20;15(14):3688. doi: 10.3390/cancers15143688. PMID 37509349

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Arm: After the gross solid tumor is removed, cold plasma is sprayed in the area of the resected tumor margins.
  Canady Helios Cold Plasma Scalpel: Device used to distribute cold plasma energy at the resected tumor margins.
  Post-operatively, patients will be started back on Adjuvant chemotherapy, radiation, or immuno-therapy as per medical oncology and multi-disciplinary team.
Period: Overall Study
Arm/Group | Primary Arm
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: The population was split between 2 institutional medical centers. The study was started in Israel, and completed in the United States.
  Participants
    United States: number analyzed (Participants) | 15
    United States | 15
    Israel: number analyzed (Participants) | 5
    Israel | 5
Tumor Type [Count of Participants; unit: Participants]
  Metastatic Recurrent Colon Cancer | 1
  Metastatic Recurrent Ovarian Cancer | 1
  Metastatic Recurrent Anal Squamous Carcinoma to the Liver (HPV Related) | 1
  Metastatic Recurrent Mesothelioma to the abdominal wall | 1
  Metastatic Recurrent Colon Cancer to the retroperitoneum | 1
  Metastatic Recurrent Myxofibrosarcoma to the chest wall | 1
  Metastatic Recurrent Breast Carcinoma to the right hip | 1
  Metastatic Recurrent Non-Small cell lung Adenocarcinoma to the left/hip/upper end of femur | 1
  Metastatic Renal Cell Carcinoma to the left clavicle | 1
  Metastatic Cholangiocarcinoma to the left elbow/distal humerus | 1
  Metastatic Non-Small Cell Lung Carcinoma (NSCLC) to right hip | 1
  Metastatic Pleomorphic Sarcoma to the left distal femur | 1
  Metastatic Recurrent Chordoma to the right gluteal posterior thigh | 1
  Metastatic Recurrent Melanoma to the left pelvis | 1
  Metastatic Pleomorphic Spindle Cell Sarcoma to the humerus | 1
  Metastatic Recurrent Squamous Cell Carcinoma to the left hand and left axillary lymph node | 1
  Metastatic Angiosarcoma of the right breast to the contralateral left breast and axilla | 1
  Metastatic Recurrent Non-Small Cell Lung Carcinoma (NSCLC) to the left hemipelvis | 1
  Metastatic Desmoplastic Small Round Cell Sarcoma (DSRCS) of left inguinal lymph node and testicle | 1
  Metastatic Recurrent Adenoid Cystic Carcinoma of the neck | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complications Due To Cold Plasma Application
Description: Adverse events (CTCAE event version 4.03 to 5.0) within 30 days after Canady Helios Cold Plasma Scalpel treatment.
Time Frame: Immediate after application of cold plasma, followed by 3 months, 6 months, 12 months and 15 month observations.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Arm
Number analyzed (Participants) | 20
Participants
  Number of participants with complications secondary to cold plasma application | 0
  Number of patients receiving cold plasma application. | 20

ADVERSE EVENTS:
Time Frame: Data has been collected for 16 months as of 5/21/21
Description: There have been 0 adverse events.
Groups:
- Primary Arm: Patients received previous chemotherapy, radiation, immuno-therapy and/or surgery prior to metastatic recurrent disease. In this study, the patients gross solid tumor was removed, and cold plasma was sprayed in the area of the resected tumor margins.
  Canady Helios Cold Plasma Scalpel: Device used to distribute cold plasma energy at the resected tumor margins.
  Post-operatively, patients will be started back on Adjuvant chemotherapy, radiation, or immuno-therapy as per medical oncology and multi-disciplinary team.
Arm/Group | Primary Arm
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Coronavirus Disease 2019 (COVID-19) global pandemic prolonged the duration of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT04267575/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT04267575/ICF_001.pdf